CLINICAL TRIAL: NCT02434367
Title: Phase 2 Randomized Study of a Walking Intervention for Radiation-related Fatigue Among Breast Cancer Patients Receiving Adjuvant Radiation
Brief Title: The Effect of Walking on Fatigue During Radiotherapy in Breast Cancer Patients 65 and Older
Acronym: WWE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The West Clinic, Memphis (Industry)
Collaborators: University of Tennessee West Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: LCCC 1412
Record Dates: First submitted 2015-04-20; First posted 2015-05-05 (Estimated); Last update posted 2017-12-14 (Actual); Status verified 2016-11

CONDITIONS: Breast Cancer; Fatigue
Keywords: Cancer
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Neoplasms | interventions — Walking

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Women randomized to the WWE program will receive a workbook, and a daily walking log, the latter to be completed during the study.
  Interventions: Behavioral: Walk With Ease Arm A
- Arm B (No Intervention): Patients randomized to the usual care arm will receive a document with information on exercise to improve fatigue during radiotherapy

INTERVENTIONS:
Behavioral: Walk With Ease Arm A — Walk With Ease is the Arthritis Foundation's evidence-based walking intervention to help with fatigue and pain. The interention is a self directed program that helps guide participants in a safe and comfortable paced walking program with an ultimate goal of walking for 30 minutes per day, five days per week.
  Other Names: WWE
  Arms: Arm A

SUMMARY:
This multicenter randomized (1:1) phase 2 study is designed to assess the efficacy of the Walk with Ease exercise program on improving fatigue after adjuvant radiotherapy compared to usual care in 50 women with stage 0-3 breast cancer who have undergone breast surgery.

Prior to initiation of radiation, during the last week, and 4-6 weeks post radiation, women in both arms will complete a number of surveys including questionnaires on fatigue, pain, depression, sleep, and social support. In addition, a blood sample will be collected prior to, during the last week of radiation, and 4-6 weeks post radiation to explore measures of inflammatory biomarkers, and their potential association with exercise and fatigue.

DETAILED DESCRIPTION:
Recruitment, consent, and randomization will occur at first postoperative visit with a radiation oncologist. A 1:1 randomization will occur between WWE program and usual care (scripted discussion on benefit of exercise during radiotherapy). Prior to initiation of radiation, women in both arms will complete 68 questions from questionnaires on pain, depression, sleep, and social support. In addition, peripheral blood will be drawn for analysis of pre-radiation measures of inflammatory biomarkers. Women randomized to the WWE program will also receive a daily walking log that they will be asked to fill out and return on the last week of radiation (6 weeks for standard fractionation and 4.5 weeks for hypofractionation), and at 4-6 weeks post radiotherapy. Also, on their last week of radiotherapy and 4-6 weeks after radiotherapy all patients will repeat the questionnaires and a blood draw for measures of inflammatory biomarkers.

Contact with study participants will be at 3 points in time after enrollment and randomization:

Baseline: At this meeting, requirements of the study will be reviewed, and study materials provided (for control arm: a one page explanation discussing the potential benefits of exercise on fatigue, for experimental arm: WWE workbook, and printed walking log). Participants will complete questionnaires and undergo other assessments including a blood draw. For those on the experimental arm, they will be asked to begin the walking program within a week, noting their walking experience in their daily log.

Last week of radiation: All participants will repeat questionnaires and other assessments during any day of their last week of radiation. A repeat blood draw will be taken. In addition those on the WWE arm will have their walking log reviewed. For those receiving hypofractionated radiotherapy, this will occur at week 4. For those receiving standard fractionation this will occur at week 6.

4-6 weeks following end of radiation: All participants will repeat questionnaires and other assessments. A repeat blood draw will be taken. In addition those on the WWE arm will have their walking log reviewed.

Patients randomized to the usual care arm will receive a document with information on exercise to improve fatigue during radiotherapy. The sheet will summarize the findings of the 3 randomized studies on exercise intervention during radiotherapy.

The primary activity required of study subjects is a 4-6-week self-directed (non-group) WWE walking program that participants do at a place and time that is convenient for them. Participants are asked to walk at a safe and comfortable pace, increasing their minutes per day at a rate they can sustain, with the ultimate goal of 30 minutes/day for at least 5 days/week. They are asked to maintain a daily walking log that is provided to them, entering total minutes per day.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years of age
* Histologically confirmed Stage I, II or III breast cancer status post breast surgery with or without adjuvant chemotherapy.
* Scheduled to undergo hypofractionated or standard fractionated radiation therapy to the breast or chest wall.
* English speaking.
* IRB approved, signed written informed consent.
* Approval from their treating radiation oncologist to engage in moderate-intensity physical activity. This will be obtained by the study research coordinator and documented on the study screening form (attached).
* Patient-assessed ability to walk and engage in moderate physical activity Willing and able to meet all study requirements.

Exclusion Criteria:

* One or more significant medical conditions that in the physician's judgment preclude participation in the walking intervention.
* Receiving accelerated partial breast irradiation.
* Unable to walk or engage in moderate-intensity physical activity.
* Already participated in Walk with Ease Program.
* Already actively walking (≥120 minutes per week).

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Compare the change in treatment related fatigue from baseline to last week of radiotherapy between patients in the WWE intervention and usual care arms using the Fatigue Symptom Index (FSI). | Four months
  change in fatigue index

SECONDARY OUTCOMES:
Compare the change in treatment related fatigue from baseline to 1-4 months post-radiotherapy between patients in the WWE intervention and usual care arms using the FSI. | Four months
  change in fatigue index
Change in Treatment Related Fatigue Symptom Index | Four months
  Compare the change in treatment related fatigue from baseline to last week of radiotherapy and to 1-4 months post-radiotherapy between patients in the WWE intervention and usual care arms using the PROMIS Fatigue 8a scale.
Change in Physical Funcionality Index | Four months
  Compare the change in physical functionality from baseline to last week of radiotherapy and to 1-4 months post-radiotherapy between patients in the WWE intervention and usual care arms using the Short Physical Performance Battery and PROMIS Short Form v1.0

OTHER OUTCOMES:
Change in Pro-Inflammatory Cytokines | Four months
  Explore the association between pro-inflammatory cytokines (TNF-α, IL-1β, and IL-6) at baseline, last week of radiation, and 1-4 months after radiation and changes in fatigue and exercise during those time periods. We will assess both the association of cycle.
Compare the change in fatigue-related side effects from baseline to last week of radiotherapy and to 1-4 months post-radiotherapy between patients in the WWE intervention and usual care arms. | Four months
  change in fatigue index
Explore the association between the change in fatigue-related side effects from baseline to last week of radiotherapy and to 1-4 months post-radiotherapy with the change in fatigue at the same time-points. | Four months
  change in fatigue index

CONTACTS AND LOCATIONS:
Overall Officials: Noam VanderWalde, MD, Principal Investigator — The West Clinic/University of Tennessee West Cancer Center
Locations (2):
- United States (2):
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - The West Clinic/ University of Tennesee West Cancer Center, Memphis, Tennessee